CLINICAL TRIAL: NCT01507064
Title: Randomized Controlled Phase II Trial Of Neoadjuvant Sorafenib Therapy Prior to Thermal Ablation for Hepatocellular Carcinoma More Than 4 cm in Size
Brief Title: Neoadjuvant Sorafenib Therapy Prior to Laser Ablation for Hepatocellular Carcinoma
Acronym: LANEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cardarelli Hospital (Other)
Responsible Party: Principal Investigator, Giovan Giuseppe Di Costanzo, Head of Hepatology, Cardarelli Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: epatologia2
Record Dates: First submitted 2012-01-05; First posted 2012-01-10 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; sorafenib; laser ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Patients who undergo to LA without sorafenib pretreatment
  Interventions: Procedure: laser ablation (LA)
- Group B (Experimental): Patients who are treated with sorafenib before LA
  Interventions: Drug: Sorafenib; Procedure: laser ablation (LA)

INTERVENTIONS:
Drug: Sorafenib — tablets 200mg dosage: 400mg bid duration: 4 weeks
  Other Names: Nexavar
  Arms: Group B
Procedure: laser ablation (LA) — For LA, we use a commercially available system (Echolaser XVG system, Esaote El.En., Florence, Italy) and four optical fibers,inserted into the tumor through four 21-gauge needles. The tips of the needles will be positioned at a distance of 15mm from each other.
  When, after LA treatments, CT or MRI findings show a residual nodule activity of 10% or less, percutaneous ethanol injection may be done. If the residual activity is of 50% or more transarterial chemoembolization may be used.

SUMMARY:
The purpose of this study is to determine whether neoadiuvant therapy with sorafenib increases the efficacy of thermal ablation in inducing the necrosis of hepatocellular carcinoma.

DETAILED DESCRIPTION:
BACKGROUND AND AIM Image-guided laser ablation (LA), minimally invasive procedure, is a potentially viable treatment option for achieving focal thermal destruction of hepatocellular carcinoma (HCC) that cannot be treated with surgery. Both techniques are effective for the destruction of small (<3 cm) tumors, but the success rate for index tumors larger than 4 cm in diameter is lower. A cause of the difficulty in treating larger tumors is represented by the heat-sink effect of tumor blood flow that limits the size of tumor ablation by drawing heat away from the tumor nodule. Surgical (Pringle maneuver) and endovascular (transarterial chemoembolization) techniques have been used to reduce the tumor blood flow during or before thermal ablation, but these techniques require invasive procedures that may decrease the patient acceptance and increase the risk of complications. Sorafenib is a multikinase inhibitor that has been approved for the treatment of advanced HCC. One of the main effect of this drug is to block vascular endothelial growth factor (VEGF) pathway, Flt-3, c-KIT, and fibroblast growth factor receptor 1, that have been shown to mediate tumor angiogenesis, reducing intratumoral blood flow. An experimental study in mice with renal cell carcinoma implanted subcutaneously, showed that treatment with sorafenib before ablation resulted in markedly decreased cancer microvessel density and significantly larger zones of radiofrequency-induced coagulation necrosis (1).

The purpose of this study is to determine if sorafenib improves the effectiveness of laser ablation (LA) for the treatment of HCC larger than 4cm in size.

1. Hakimé A, Hines-Peralta A, Peddi H, Atkins MB, Sukhatme VP, Signoretti S, Regan M, Goldberg SN. Combination of Radiofrequency Ablation with Antiangiogenic Therapy for Tumor Ablation Efficacy: Study in Mice. Radiology 2007, 244, 464-470.

STUDY DESIGN

Participants will be randomized to receive either sorafenib (400mg twice a day) or placebo continuously for 4 weeks (on days 1-28). LA will be performed on day 29. On days 0 and 28, and 1, 6, and 12 months after LA, patients will undergo to a physical exam. Adverse events will be recorded using a pre-planned questionnaire in accordance with the "common toxicity criteria".

Occurrence and characteristics of postablation syndrome will also be recorded. During a six-month period, if clinically indicated LA procedures preceded by a four-week sorafenib treatment, may be repeated up to three times.

Laboratory values will be assessed on days 0 and 28, and 1, 6, and 12 months after the first LA procedure.

Upper gastrointestinal endoscopy will be done before starting drug treatment. A tumor biopsy will be obtained at the time of the first LA. A CT or MRI scan will be performed at the time of inclusion in the study, at 1, 6, and 12 months after LA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* ECOG = 0 or 1
* No liver decompensation (Child-Pugh <8), bilirubin <3mg/dL
* Patients with unresectable HCC or who refused surgery
* Confirmed HCC by pathology or by AASLD imaging guidelines
* At least one HCC nodule (index tumor) accurately measured as 4-8cm in diameter on baseline imaging
* No prior therapy for the index tumor
* No prior systemic treatment for HCC within 4 weeks of study entry
* LA clinically indicated for index tumor
* Hemoglobin >9.0 g/dl; Platelet count correctable to >50,000/mm3; INR correctable to <2.0.

Exclusion Criteria:

* Other severe concomitant diseases that may reduce life expectancy
* Participants currently receiving any other study agents
* Cancer vascular invasion or extrahepatic metastasis
* Uncontrolled hypertension
* Thrombotic events or myocardial infarction within the past 6 months
* Hemorrhage/bleeding event within 4 weeks
* Evidence of severe or uncorrectable bleeding diathesis or coagulopathy
* Contraindication to or inability to undergo the LA procedure
* Human immunodeficiency virus (HIV) infection
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Effectiveness of sorafenib in increasing the effectiveness of laser ablation (LA) | 1 year
  Measures: complete tumor ablation rate (according to the mRECIST), time-to-recurrence (in complete response subgroup), time-to-progression (in partial response subgroup).

SECONDARY OUTCOMES:
Safety of sorafenib treatment prior to LA. | 6 months
  Measure: incidence and grade of adverse events in patients treated with sorafenib (group B)
Survival in the two treatment groups | 2 years
  Measured from the date of LA until the date of death or last visit

CONTACTS AND LOCATIONS:
Locations (1):
- UOSC Epatologia - Cardarelli Hospital, Napoli, Italy